CLINICAL TRIAL: NCT05487638
Title: The Effect of Telephone Nursing Education and Counseling Services Given to Patients With Coronary Artery Bypass Graft on Discharge Satisfaction Level and Self-Care Strength of Patients: A Randomized Controlled Study
Brief Title: The Effect of Telephone Nursing Education and Counseling Services Given to Satisfaction Level and Self-Care Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Vesile Eskici Ilgin, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: vesile2022
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Complications
Keywords: surgical site infection; coronary artery bypass graft; constipation; sleep disorders; pain
MeSH Terms: conditions — Postoperative Complications; Surgical Wound Infection; Constipation; Sleep Wake Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental Group (Experimental): Training was given to the patients once a week, starting on the second day after discharge, four times in total. Increasing the level of knowledge about infection control, wound care, post-CABG care, using drugs as prescribed, hygiene, excretion (things to be done to avoid constipation), nutrition (diet and diet compliance after CABG), bleeding control, proper sleep and rest positions, deep breathing and coughing exercises, maintaining a healthy weight, what to pay attention to while taking a bath, pain management and methods of coping with pain, relaxation techniques, walking and exercise, returning to social life, reducing anxiety and depression, using elastic stockings and chest corsets, controlling Training was given on the subjects of notifying the due dates, emotional adjustment and coping methods with symptoms. After 1 month of training, at the end of the 4th week, the patients were asked to fill out the Discharge Education Satisfaction Scale and the Self-Care Strength Scale.
  Interventions: Other: Nursing Education and Counseling Service Provided to Patients by Video Calling on the Phone
- Control Group (No Intervention): On the other hand, no intervention was made in the control group and after discharge, the personal information form, the Discharge Training Satisfaction Scale and the Self-Care Strength Scale were filled. At the end of the 4th week, the patients were asked to fill out the Discharge Education Satisfaction Scale and the Self-Care Strength Scale.

INTERVENTIONS:
Other: Nursing Education and Counseling Service Provided to Patients by Video Calling on the Phone — Nursing Education and Counseling Services were provided to the patients by video calling on the phone for the problems they may encounter in the postoperative period.
  Other Names: İntervention Group
  Arms: experimental Group

SUMMARY:
In the post-discharge period, it is important to follow the patients from home by telephone and to provide the necessary nursing education and counseling services, increasing the self-care powers of the patients, increasing their quality of life, adapting to the social life after discharge and facilitating the patient's adaptation to the post-discharge process.

When the literature is examined, it can be said that the study is original since there are no studies on this subject. The aim of this study is to determine the effect of nursing education and counseling service given to patients who have undergone CABG, on the level of discharge satisfaction and self-care power of patients.

DETAILED DESCRIPTION:
Cardiovascular diseases are one of the leading causes of death globally, with an alarming prevalence. The World Health Organization (WHO) stated that 17.9 million people died from cardiovascular diseases in 2019, and this number constituted 32% of the death rates worldwide At the same time, it is emphasized that 14.2% of all deaths by 2030 may be caused by coronary heart diseases There are multiple approaches to the treatment of coronary heart diseases. Healthy lifestyle behaviors form the basis of these approaches. However, in cases where these approaches are not sufficient, surgical treatment is required. In this case, one of the surgical procedures applied is Coronary Artery Bypass Graft (CABG). CABG procedure is a risky and important surgical procedure applied all over the world After CABG, life-threatening complications can be seen after CABG due to reasons such as sternotomy wound, ventilator support lasting 12-24 hours after surgery, hospital stay of 5-10 days on average, and recovery period lasting 6-8 weeks.

In a study, it is stated that more than 200,000 CABG surgeries are performed annually in the United States, and approximately 14% of these patients present to the emergency department with postoperative complications within 30 days of discharge. The golden rule in centers where cardiac surgery is performed in England is the patient's 6-7th postoperative day. day discharge. However, 6-7 days after surgery. It has been reported that the patient's sternotomy wound has not fully healed on the same day, and life-threatening complications may occur if appropriate care is not provided. It is possible to prevent these complications or to ensure their early diagnosis with good nursing care. Good nursing care includes a planned discharge training.

Today, the purpose of health services; In addition to prolonging the life span, it is to help the individual cope with his problems, to increase his self-care power and self-efficacy perception, to improve his independence and quality of life by strengthening his knowledge and skills. Quality/effective care and education to be applied by healthcare professionals to the patient and their relatives undergoing CABG; It plays an important role in preventing repeated hospitalizations, increasing self-care power and self-confidence, and gaining independence of the patient.

Self-care is the continuous participation of an adult in activities aimed at maintaining and maintaining their own health and well-being. Self-care disability occurs when there is an imbalance between caring power and the need for therapeutic self-care. When there is an imbalance between the individual's self-care abilities and needs, the need for nursing intervention arises. Investigation of Self-Care Behaviors in Patients with Chronic Heart Failure After CABG surgery, in addition to physical problems such as pain in the incision area in the chest or leg, weight loss, respiratory distress, sleep disorders, fatigue, exhaustion, loss of appetite, constipation, difficulty in bathing and limitation of body movements, unhappiness, difficulties in coping with stress, Psychosocial problems such as anxiety, even depression, role complexity in the family, decrease in physical activities, changes in work life, changes in social relations and sexual life are observed. These physical and psychosocial problems reduce the self-care power of patients. In the studies, while the surgical patients were discharged, the most; It has been determined that they need information about incision/wound care, pain control, activities of daily living, drug use, possible complications and excretion. In the study of Yılmaz and Çiftçi, it was found that all of the patients experienced activity, 95.6% nutrition, 88.9% sleep and 86.7% excretion problems within a week after discharge.

The nurse has an important role in preparing the patient and family of patients undergoing surgery for discharge and helping them to accept the current situation. Within the scope of discharge planning, the nurse should provide information that can help patients increase their self-care power at home after discharge, adapt to the new situation and prevent possible complications. In the studies conducted, the patients who were given discharge training; It is stated that the recovery processes accelerate, their self-confidence increases in parallel with their self-care abilities, the number of repeated admissions to the hospital/outpatient clinic decreases, and accordingly, patient care costs decrease and the quality of care increases.

In the post-discharge period, it is important to follow the patients from home by telephone and to provide the necessary nursing education and counseling services, increasing the self-care powers of the patients, increasing their quality of life, adapting to the social life after discharge and facilitating the patient's adaptation to the post-discharge process.

When the literature is examined, it can be said that the study is original since there are no studies on this subject. The aim of this study is to determine the effect of nursing education and counseling service given to patients who have undergone CABG, on the level of discharge satisfaction and self-care power of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient between the ages of 18 and 75,
* literate, who could speak Turkish,
* who had undergone CABG surgery for the first time,
* who could be contacted,
* who did not have a mental illness,
* whose discharge was decided,
* who stayed in the hospital for at least 2 nights after the operation,
* who voluntarily agreed to participate in the study were included.

Exclusion Criteria:

* patients whose surgery was delayed
* Patients who refused to participate in the study
* developing mental problems
* patients whose discharge was canceled

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Discharge Training Satisfaction Scale star_border Discharge Training Satisfaction Scale | up to 1 month
  Discharge Education Satisfaction Scale is in five-point Likert type (from 1 to 5): 3 items about discharge process, 3 items about personal information, 7 items about home care, 3 items about infection, 5 items about controls, It consists of 21 questions in total.
Self-Care Strength Scale | up to 1 month
  It was adapted into Turkish by Nakhchivan N. This scale consists of 43 descriptive statements. Each statement was scored from 0 to 4 in the 5-point Likert-type Self-Care Scale. Scoring of the scale items is (0) does not describe me at all, (1) does not describe me very well, (2) I have no idea, (3) describes me a little, (4) describes me a lot. It describes the self-care powers of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Vesile Eskici İlgin, Dr, Principal Investigator — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Palandöken, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No